CLINICAL TRIAL: NCT06407674
Title: Non-invasive Assessment of RECTUM (POUCH) by US (RECT-US): Multicentric, Observational and Cross-sectional Comparison Study With Colonoscopy in a Cohort of IBD Patients
Brief Title: Non-invasive Assessment of RECTUM (POUCH) by US (RECT-US) in a Cohort of IBD Patients
Acronym: RECT-US
Status: Recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Mariangela Allocca, M.D, PhD, IRCCS San Raffaele
Other Study IDs: RECT-US
Record Dates: First submitted 2024-05-06; First posted 2024-05-09 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Ulcerative Colitis; Crohn's Disease
Keywords: intestinal ultrasound; Ileocolonoscopy; Trans-perineal ultrasound
MeSH Terms: conditions — Colitis, Ulcerative; Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ulcerative colitis
- crohn's disease

SUMMARY:
At enrollment, after informed consent form will be discussed and signed, subjects will undergo complete disease assessment.

In this study, 150 adult subjects with IBD will be enrolled at the Gastroenterology Department of the San Raffaele Hospital (50 patients with Crohn's disease, 50 with Ulcerative colitis not undergoing proctocolectomy, and 50 with Ulcerative colitis undergoing proctocolectomy with ileal pouch-anal anastomosis).

All the patients will perform routine investigations with Ileocolonoscopy (IC), according to the current standard of care indications and ECCO guidelines, and they will be assessed by both Intestinal Ultrasound (IUS) and Trans-perineal ultrasound (TPUS). Blood and stool samples will be obtained for fecal calprotectin (FC) and C-reactive protein (CRP) measurements, respectively, as normal clinical practice.

All the procedures of this study are performed routinely in clinical practice. All the procedures are performed in a single day-visit for the patient.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of IBD for at least 3 months, in particular 50 with Crohn&;s disease (CD), 50 with ulcerative colitis (UC) not undergoing proctocolectomy, 50 with ulcerative colitis (UC) undergoing proctocolectomy with ileal pouch-anal anastomosis
* Performing ileocolonoscopy, according to current standards of care and ECCO guidelines, will be assessed by both IUS and TPUS. Procedures performed routinely in clinical practice
* Ability to understand and comply with the study procedure and sign an informed consent form

Exclusion Criteria:

* Pregnancy;
* Concomitant intestinal infection (e.g. Clostridium difficile);
* Cirrhosis or intra-abdominal ascites.
* Subjects not able to comply with any study procedure;
* Subjects not able to understand and give informed consent form;
* Subjects with any contraindication to any study procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 150 adult subjects (minimum age: 18 years) with IBD (established diagnosis since at least 3 months), specifically 50 with CD, 50 with UC not undergoing proctocolectomy, 50 with UC undergoing proctocolectomy with ileal pouch-anal anastomosis, irrespective of concomitant therapy, performing routine investigations with IC, according to the current standard of care indications and ECCO guidelines, will be assessed by both IUS and TPUS. Procedures performed routinely in clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-01-10 (Actual); Primary Completion 2024-11-28 (Estimated); Study Completion 2025-05-28 (Estimated)

PRIMARY OUTCOMES:
correlation of data | 1 day (Cross Sectional study)
  To correlate ultrasound finding, both transabdominally and transperineally, with endoscopic findings

CONTACTS AND LOCATIONS:
Locations (1):
- Irccs San Rafael Hospital, Milan, Italy